CLINICAL TRIAL: NCT05587972
Title: Real World Treatment Experience of Patients With Breast, Lung, or GI Cancer or Multiple Myeloma Using Remote Symptom Monitoring
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPT-IN Research Protocol
Record Dates: First submitted 2022-10-07; First posted 2022-10-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Lung Cancer; Gastrointestinal Cancer; Multiple Myeloma
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms; Multiple Myeloma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — Patients will complete a baseline survey in person using a secured device or remotely using their own electronic device in a location of their choice. Weekly electronic PRO surveys are collected from the patients using the Carevive platform for a minimum of 12 weeks.

SUMMARY:
The Carevive registry collects patient characteristics, patient symptoms, and treatment experience data from patients receiving cancer treatment for breast, lung, GI or multiple myeloma. For this study, a core set of variables is collected on each patient in the Carevive platform. Patients will complete a baseline survey in person using a secured device or remotely using their own electronic device in a location of their choice. Weekly electronic Patient Reported Outcome surveys are collected from the patients using the Carevive platform for a minimum of 12 weeks. Patients may continue weekly surveys as long as they are receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years of age or older.
* Subjects may be any stage and anywhere in the treatment continuum.
* Subject participants must have a diagnosis of breast, lung, GI or ovarian cancer or multiple myeloma.
* Subjects must be able to complete on-line surveys using a cell phone, tablet, or computer.
* All participants must be able to understand English.

Exclusion Criteria:

* Any patient who cannot understand written or spoken English.
* Any patient without the ability to complete on-line surveys using a cell phone, tablet, or computer.
* Any patient on a treatment clinical trial.
* Any prisoner and/or other vulnerable persons as defined by NIH (45 CFR 46, Subpart B, C and D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-10-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Create data set | 12 weeks
  Project outcome measures for this project are the prevalence, frequency, and severity of symptoms in each disease group, longitudinal change in symptom experience, and time on treatment from enrollment to next treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Galaznik, MD, Study Director — Carevive Systems, Inc.
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No